CLINICAL TRIAL: NCT03057236
Title: A Pilot Feasibility Study of a Cognitive Behavioral Coping Skills (CBCS) Group Intervention for Patients Undergoing Antiviral Therapy for Chronic Hepatitis C
Brief Title: Pilot Feasibility Study of a Cognitive Behavioral Coping Skills (CBCS) Group Intervention for Hep C Therapy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-2323; K23DK089004 (NIH); K24DK066144 (NIH)
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis C; Hepatitis C, Chronic
Keywords: psychological, behavioral, psychosocial, antiviral, liver
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Behavior

STUDY DESIGN:
Intervention Model Description: Participants are assigned to Standard of Care group or the Intervention (CBCS) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): This arm does not receive the behavioral intervention. Participants will complete HCV treatment per standard of care.
- Cognitive Behavior Coping Skills (Experimental): The CBCS intervention is a structured module-based group intervention involving 9, 2-hour sessions. Participants will participate in 4 weekly sessions before HCV treatment to learn and practice new cognitive behavioral skills, and 5 sessions during HCV treatment at weeks 2, 4, 6, 8, and 12.
  Interventions: Behavioral: Cognitive Behavior Coping Skills

INTERVENTIONS:
Behavioral: Cognitive Behavior Coping Skills — The CBCS-HCV is a psychosocial intervention delivered in group format. Through 9 group sessions, patients will learn coping skills, relaxation techniques and other new cognitive and behavioral skills based on several empirically-supported cognitive behavioral interventions.
  Other Names: CBCS-HCV
  Arms: Cognitive Behavior Coping Skills

SUMMARY:
This is a pilot feasibility study of a small randomized controlled trial (RCT)design to evaluate participation in a Cognitive Behavioral Coping Skills (CBCS) group intervention versus standard of care in patients with hepatitis C undergoing antiviral treatment. The primary objectives are to (1) examine effect size (ES) estimates of key outcomes to provide essential data to inform a larger efficacy trial, (2) determine whether clinically significant improvements occurred in any key outcomes, and (3) evaluate study feasibility and patient acceptability. Study findings will inform a larger efficacy study of the CBCS-HCV.

DETAILED DESCRIPTION:
This is a pilot feasibility study of a Cognitive Behavioral Coping Skills (CBCS) Group Intervention with a representative sample of patients with Hepatitis C viral (HCV)undergoing standard antiviral treatment in a small RCT to examine (1) study feasibility, (2) effect size estimates, and (3) whether clinically significant improvements occurred in key outcomes. This pilot study will allow the investigators to test the hypotheses that the study procedures are feasible and that participation in the CBCS-HCV group is acceptable and useful to participants. Furthermore, effect size estimates of key outcome variables will determine which outcomes appear to improve as a result of the intervention and should potentially be evaluated in a future efficacy study. Several patient-reported outcomes (PROs) are evaluated: health-related quality of life (HrQOL), perceived stress, depression, anxiety, anger, fatigue, sleep, pain and medication adherence. The investigators will also determine if group participation affects viral cure rate. Change scores that have an effect size d> .35 are considered potentially clinically significant and reasonable to evaluate in a larger efficacy study. Study feasibility elements evaluated included: feasibility of a RCT study design, intervention delivery, patient acceptability, therapist protocol fidelity, recruitment, enrollment, attendance, retention and data collection.

The investigators planned to enroll and evaluate the intervention in two waves of study participants (Wave 2, Wave 3). When a block of 12 patients is consented for Wave 2, participants will be randomized to standard of care (SC; n=6) or the CBCS-HCV group intervention (n=6). The same procedure will be used to consent and randomize 12 patients in Wave 3 to SC vs CBCS-HCV. Patients randomized to CBCS will participate in 4 weekly CBCS sessions prior to starting HCV treatment, and 5 more sessions during HCV treatment, on the same day they attend follow-up treatment visits at weeks 2, 4, 6, 8, and 12. Outcome data will be collected at baseline (T1), just prior to HCV treatment starting (T2); at week 8 of HCV treatment (T3), at end of CBCS intervention/ HCV treatment at week 12 (T4), and 1-month post-CBCS intervention/ HCV treatment (T5). The primary outcome is change in total HrQOL score. Secondary outcomes are change in other PROs noted above. Additional secondary outcomes are group differences in medication adherence and viral cure rate. Elements of study feasibility are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All English -speaking adult patients (age 21 or older) with HCV;
* Treatment-naïve or treatment experienced;
* Deemed eligible for standard antiviral therapy for HCV by the clinical providers by standard clinical criteria;
* Referred by HCV clinician or on "Treatment Waitlist" ready to start a 12-week prescribed course of antiviral therapy.

Exclusion Criteria:

* Prescribed a 24-week antiviral treatment regimen;
* Inability to provide written informed consent;
* Currently participating in another pharmaceutical clinical trial of hepatitis C therapeutics;
* Evidence of use of illicit substances (excluding marijuana) reported in the last 6 months by patient during screening or noted in patient's medical record
* Current significant suicidal ideation reported during Screening or noted in patient's medical record
* Current significant personality disorder or features reported during Screening or noted in patient's medical record that is clinically judged to be detrimental to the group therapeutic setting for other group participants
* Cannot make personal commitment to attend study visits and/or intervention sessions
* Is medically or psychiatrically contraindicated to proceed with HCV antiviral therapy at the time of study enrollment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Change in health related quality of life score from T1 to T2 | 4 weeks
  HRQOL is measured using the Functional Assessment of Cancer Therapy-General Population (FACT-GP). The FACT-GP is an instrument derived from the Functional Assessment of Chronic Illness Therapy (FACIT) measurement system to measure HRQOL during the management of chronic illness. The FACT-GP is a 21-item survey that assesses four HRQOL domains: Physical well-being; Social/Family well-being; Emotional well-being; and Functional well-being. Items are rated on a five-category response system ranging from 0 (not at all) to 4 (very much). Higher scores indicate higher (better) HRQOL. Change in the total HRQOL score from T1 to T2 was the primary outcome measure, with an effect size d>.35 indicating a small to moderate clinical improvement

SECONDARY OUTCOMES:
Change in 4 HRQOL subscale scores (physical well-being, emotional well-being, social well-being, functional well-being) from T1 to T5 | 20 weeks
  Change in each of the 4 HRQOL subscale scores derived from the FACIT-GP will be evaluated. Items are rated on a five-point system ranging from 0 (not at all) to 4 (very much). Higher scores indicate higher (better) physical, emotional, social, and functional well-being. Change in these 4 subscale scores from T1 to T5 evaluates change from baseline to 1 month post-intervention/post-HCV treatment. An effect size change of d>.35 would indicate a small to moderate clinical improvement
Change in 4 HRQOL subscale scores (physical well-being, emotional well-being, social well-being, functional well-being) from T1 to T2 | 4 weeks
  Change in each of the 4 HRQOL subscale scores derived from the FACIT-GP will be evaluated. Items are rated on a five-point system ranging from 0 (not at all) to 4 (very much). Higher scores indicate higher (better) physical, emotional, social, and functional well-being. Change in these 4 subscale scores from T1 to T2 evaluates change after 4 CBCS sessions. An effect size change of d>.35 would indicate a small to moderate clinical improvement
Change in perceived stress scale score from T1 to T2 | 4 weeks
  The Perceived Stress Scale (PSS) is a widely used survey to measure stress perception. The scale includes 10 items, rated using a 5-point Likert scale, from 0 (never) to 4 (very often) where patients report the frequency of symptoms in the past month. The PSS has been shown to have good reliability and validity. Higher stress scores represent a worse outcome. T1 to T2 measures change after 4 CBCS sessions. An effect size change of d>.35 indicates a small to moderate clinical improvement
Change in perceived stress scale score from T1 to T5 | 20 weeks
  The Perceived Stress Scale (PSS) is a widely used survey to measure stress perception. The scale includes 10 items, rated using a 5-point Likert scale, from 0 (never) to 4 (very often) where patients report the frequency of symptoms in the past month. The PSS has been shown to have good reliability and validity. Higher stress scores represent a worse outcome. T1 to T5 measures change from baseline to 1 month post-intervention/post HCV treatment. An effect size change of d>.35 indicates a small to moderate clinical improvement
Change in 8 PROMIS symptom scores from T1 to T2 | 4 weeks
  PROMIS symptom surveys measured 8 constructs: depression, anxiety, anger, fatigue, pain, sleep disturbance, sleep impairment, pain intensity, and pain interference. These surveys utilize 4-8 items each with higher scores indicating higher (worse) symptoms. The PROMIS surveys are derived from the Patient-Reported Outcome Measurement Information System (PROMIS). Responses are scored 1 to 5 for each item with higher scores representing worse outcomes. Raw total scores are translated into T-scores in which the raw score has been rescaled into a standardized score with a mean of 50 and a standard deviation of 10. T1 to T2 measures change from baseline to after 4 CBCS sessions. An effect size change of d>.35 indicates a small to moderate clinical improvement
Change in 8 PROMIS symptom scores from T1 to T5 | 20 weeks
  PROMIS symptom surveys measured 8 constructs: depression, anxiety, anger, fatigue, pain, sleep disturbance, sleep impairment, pain intensity, and pain interference. These surveys utilize 4-8 items each with higher scores indicating higher (worse) symptoms. The PROMIS surveys are derived from the Patient-Reported Outcome Measurement Information System (PROMIS). Responses are scored 1 to 5 for each item with higher scores representing worse outcomes. Raw total scores are translated into T-scores in which the raw score has been rescaled into a standardized score with a mean of 50 and a standard deviation of 10. T1 to T5 measures change from baseline to 1 month post-intervention/post-HCV treatment. An effect size change of d>.35 indicates a small to moderate clinical improvement
Pill count medication adherence | 12 weeks
  To assess medication adherence from week 2 to 12 of HCV treatment, patients brought HCV medication bottles to clinic and pills were counted at treatment weeks 2, 4, 6, 8, and 12 if a patient had a standard clinical visit. The number of pills remaining in the pill bottle were monitored to determine ideal vs actual proportion of pills taken between clinic visits. The proportion of pills taken at each visit was added then divided by the number of visits to obtain an overall proportion of medical adherence.
Viral cure after HCV treatment | 20 weeks
  Medical records were reviewed for lab results for HCV RNA viral load after treatment had ended for at least 4 weeks. Lab data for HCV RNA indicated "detectable virus: or "undetectable virus" indicating whether viral cure had been achieved.
study feasibility 1: Feasibility of recruitment | 3 months
  Feasibility of recruitment efforts will be determined by the proportion of patients contacted for screening via phone versus those who are consented
study feasibility 2: Feasibility of randomization | 3 months
  Feasibility of randomization will be determined by whether the investigators were able to enroll and randomize a block of 12 participants for Wave 2 and Wave 3
study feasibility 3: Feasibility of enrollment | 3 months
  Feasibility of enrollment will be determined by the proportion of patients consented vs those enrolled and randomized
study feasibility 4: Feasibility of data collection | 20 weeks
  Feasibility of data collection will be determined by the overall proportion of surveys completed by each participant at each of the 5 timepoints (T1-T5)
study feasibility 5: Patient retention and acceptability | 16 weeks
  Patient acceptability of the CBCS intervention will be determined by retention, defined as the overall number of CBCS sessions attended by each patient and the proportion of patients who started and finished the intervention
Patient acceptability and comprehension | 16 weeks
  CBCS-HCV participants will complete a 14-item brief survey administered by a research coordinator at the end of each of the 9 sessions to rate the session on acceptability, usefulness, comprehension, and group process. Each item is rated on a five-point Likert scale from "1=Not At All" to "4=A lot/Extremely" with higher scores indicating greater patient acceptability. The survey was adapted from one developed by previous interventionists to examine intervention acceptability.
Therapist Competency in intervention delivery | 16 weeks
  Study staff will observe the delivery of each of the 9 CBCS module-based sessions and complete an observer-rating form of the therapist's competency. Ratings are made on 14 items based on the following Likert scale: 1=Not At All; 2=A little; 3=moderately; and 4=A lot/Extremely with higher scores indicating greater competency to manage group dynamics and demonstrate awareness of the nonspecific therapeutic processes.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Evon, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evon DM, Golin CE, Ruffin R, Ayres S, Fried MW. Novel patient-reported outcomes (PROs) used in a pilot and feasibility study of a Cognitive Behavioral Coping Skills (CBCS) group intervention for patients with chronic hepatitis C. Pilot Feasibility Stud. 2018 Jun 27;4:92. doi: 10.1186/s40814-018-0285-5. eCollection 2018. PMID 29983993